CLINICAL TRIAL: NCT06128668
Title: The Effect of Yoga on Sleep Quality, Fatigue and Physical Activity Level of Multiple Sclerosis Patients: A Randomized Controlled Study
Brief Title: The Effect of Yoga on Sleep Quality, Fatigue and Physical Activity Level of Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 338394
Record Dates: First submitted 2023-10-24; First posted 2023-11-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
Keywords: Fatigue; Sleep Quality; Yoga
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Sleep Initiation and Maintenance Disorders | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): Yoga will be aplicated
  Interventions: Behavioral: Yoga
- Control (No Intervention): Yoga will not be aplicated

INTERVENTIONS:
Behavioral: Yoga — Yoga will be applied
  Arms: Yoga

SUMMARY:
This randomized controlled study will be conducted to examine the effects of Yoga on Sleep, Fatigue and Physical Activity in Individuals Diagnosed with Relapsing-Remitting Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with Relapsing-Remitting Multiple Sclerosis Being an adult between the ages of 18-65

Exclusion Criteria:

* Those who have communication problems Those with psychiatric problems Having a condition that prevents you from doing yoga

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Six week
  A reliable distinction can be made at the desired level between "good sleepers" and "poor sleepers". The scale contains a total of 24 questions, 19 of which are self-evaluation questions. 5 of them are answered by the individual's spouse or roommate, are used only for clinical information and are not included in the scoring. Question 19, one of the self-assessment questions, is about whether there is a roommate or spouse and is not taken into account in determining the total and component scores of the scale. Scale questions that determine sleep quality include different factors related to sleep quality. These questions are to determine sleep duration, sleep latency, and the frequency and severity of specific sleep-related problems. The 18 items scored were grouped into 7 component scores.
Fatigue Severity Scale: | six week
  The Fatigue Severity Scale is used in most studies evaluating fatigue in MS. The scale consists of 9 questions. Each question consists of 7 points. High scores indicate fatigue. The validity and reliability studies of the scale for Turkey were conducted by Armutlu et al. in 2007, and the Turkish version was also found to be valid and reliable. The scales include the day they were filled in and inquire about fatigue status in the last month. The Fatigue Severity Scale was developed in the 1980s to facilitate the research and treatment of fatigue and to distinguish fatigue from depression and somatic disorders. The survey demonstrated good internal consistency when repeated and across disease responses. The validity of the questionnaire was found to be higher in MS patients.
Expanded Disability Status Scale (EDSS, ExpandedDisabilityStatusScala): | six week
  This test, created by Kurtzke, measures disability and neurological symptoms in MS patients. A score is given between 0 and 10. 0 indicates no disability or disorder, while 10 indicates death due to MS. MS patients were divided into 2 groups according to their EDSS scores. EDSS = 6 (requires cane, crutches or other aids to walk)
International Physical Activity Questionnaire (IPAQ): | six week
  It obtains data on sitting, walking, moderate-intensity activities and time spent in vigorous activities. In evaluating all activities, the criterion is that each activity should be done for at least 10 minutes at a time. A score as METmin/week is obtained by multiplying the minute, day and MET value. After scoring, physical activity levels are classified as physically inactive (inactive), low physical activity level (minimally active) and sufficient physical activity level (very active). It has short and long forms, and the short form is generally used in studies. The short form consists of 8 questions

CONTACTS AND LOCATIONS:
Locations (1):
- Gülcan Bahçecioğlu TURAN, Elâzığ, Turkey (Türkiye)